CLINICAL TRIAL: NCT06863337
Title: Glucose Pattern in Infertile Women Receiving Assisted Reproduction: a Prospective Study Using Continuous Glucose Monitoring
Brief Title: Glucose Pattern in Infertile Women Receiving Assisted Reproduction Using Continuous Glucose Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Principal Investigator, Professor, Chief Physician, Deputy Director, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20250303
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-03

CONDITIONS: Infertility Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- wearing continuous glucose monitorings (Experimental): Patients will wear two FreeStyle Libre Pro Flash CGM (Abbott Diabetes Care, Alameda, CA, USA) to ensure continuous tracking of blood glucose levels at key time points throughout the ovarian stimulation.
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Each patient will participate in the group only once and wear two FreeStyle Libre Pro Flash CGM (Abbott Diabetes Care, Alameda, CA, USA), which record glucose readings for up to 14 days.
  Following the initial consultation and before initiating the ovulation induction protocol, the first CGM sensor will be placed to collect baseline data. Upon entering the ovulation induction cycle, patients will return to the hospital on the 2nd or 3rd day of menstruation, at which point the first CGM sensor will be removed, and the second sensor will be applied. This second sensor will be removed after 14 days.
  In summary, this protocol ensures continuous tracking of blood glucose levels at key time points throughout the ovarian stimulation.

SUMMARY:
No studies have been seen on glucose variation during medication for assisted reproduction. The aim of this study is to continuously observe glucose variation during assisted reproduction treatment using continuous glucose monitoring (CGM), and to further explore whether glucose variation will affect the outcomes related to assisted reproduction.

DETAILED DESCRIPTION:
Infertility is a growing global health concern and affects approximately 20% of couples of reproductive age. As a result, the use of assisted reproductive technologies (ART) is becoming more prevalent. This study could serve as a basis for the interpretation of glucose levels with respect to these people undergoing ART regimen. Moreover, the success rate of ART still needs to be further improved. Key challenges include optimizing the hormonal components of ART regimens and determining the ideal treatment duration. This study might provide insights into the potential benefits of monitoring glucose levels at specific points during ART cycles (which is not usually performed in routine practice) and help clinicians tailor ART regimen to minimize glucose variation, ultimately improving clinical pregnancy and live birth rates. Additionally, the findings might support integrating CGM into the clinical practice of ART, enhancing individualized patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent and voluntary participation in this study;
2. Age ≥ 18 years and ≤40 years old;
3. Infertile patients who will undergo their first or second cycle of in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) at the study center;
4. The chosen ovulation promotion regimens is the GnRH antagonist regimen/progesterone-promoting ovulation under hyperprogesterone state (PPOS) regimen.

Exclusion Criteria:

1. Recent infections (excluding viral infections of the reproductive system such as HPV);
2. Recent glucocorticoid treatment or chemotherapy;
3. Clinical conditions affecting the outcome of assisted reproduction, including repeated implantation failure, recurrent spontaneous abortion, history of unilateral oophorectomy, uterine malformations, and parental karyotype abnormalities;
4. Participants were unable to tolerate tape adhesive around sensor placement area, or with medically documented allergy towards the adhesive (glue) of plasters, or with serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) around sensor placement area.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean sensor glucose (MSG) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Mean of daily continuous 24-h blood glucose

SECONDARY OUTCOMES:
time in tight range(3.9~7.8mmol/L, %) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Percentage of time within glucose level of 3.9-7.8 mmol/L (70-140 mg/dL) measured by CGM
Time below range (<3.9mmol/L, %) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Percentage of time below glucose level of 3.9 mmol/L (70 mg/dL) measured by CGM.
Time above range (>7.8mmol/L, %) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Percentage of time above glucose level of 7.8 mmol/L (140 mg/dL) measured by CGM
Coefficient of variation (CV) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Standard deviation divided by mean glucose level measured by CGM
Standard deviation (SD) | Through study completion (during assisted reproductive treatment period，about 2 months）
  Standard deviation of blood glucose measurements during CGM

OTHER OUTCOMES:
Number of oocytes retrieved | Through study completion (during assisted reproductive treatment period，about 2 months）
  The number of oocytes obtained under ultrasound guidance
Oocyte retrieval rate | Through study completion (during assisted reproductive treatment period，about 2 months）
  Oocyte Retrieval Rate = Number of Oocytes Retrieved / Number of Follicles
Number of MII oocytes | Through study completion (during assisted reproductive treatment period，about 2 months）
  The number of metaphase II oocytes that have nuclear maturity at the time of injection
Rate of MII oocytes | Through study completion (during assisted reproductive treatment period，about 2 months）
  the proportion of oocytes that have nuclear maturity at the time of injection
Rate of high-quality embryos | Through study completion (during assisted reproductive treatment period，about 2 months）
  the proportion of Day 2 and Day 3 embryos with high score or grade
Biochemical pregnancy rate | Through study completion (during assisted reproductive treatment period，about 6 months）
  The proportion of pregnancies confirmed by the detection of hCG in serum or urine, but without ultrasound confirmation of a gestational sac or fetal heartbeat.
Clinical pregnancy rate | Through study completion (during assisted reproductive treatment period，about 6 months）
  The proportion of pregnancies confirmed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy
Miscarriage rate | Through study completion, about 1 year
  The proportion of pregnancies that end spontaneously before 28 weeks of gestation after confirmation of clinical pregnancy
Live Birth Rate | Through study completion, 18 months
  The proportion of successful deliveries resulting in a live-born infant.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No